CLINICAL TRIAL: NCT00780000
Title: Phase 2 Clinical Trial of Intravenous Alvespimycin [KOS-1022] in Patients With Her2 Positive Breast Cancer
Brief Title: Clinical Trial of Intravenous Alvespimycin in Patients With Her2 Positive Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA201-002; 2007-003121-25 (EudraCT Number); KDG-201 (Other: Kosan)
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — 17-(dimethylaminoethylamino)-17-demethoxygeldanamycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A1 (Experimental)
  Interventions: Drug: Alvespimycin

INTERVENTIONS:
Drug: Alvespimycin — Solution, IV, Alvespimycin 80 mg/m2, Weekly one hour infusion Days 1, 8, and 15, every 4 weeks thereafter until disease progression or DLT

SUMMARY:
The purpose of this study is to determine the anti-tumor activity (via objective response rate) of alvespimycin in patients with breast cancer who have not previously received trastuzumab (except as adjuvant therapy).

ELIGIBILITY:
Inclusion Criteria:

* KPS performance status of >= 80% ("normal activity with effort")
* Metastatic breast cancer with Her2 amplification by FISH or 3+ Her2 overexpression by immunohistochemistry ("IHC")
* Must have received no more than one prior cytotoxic chemotherapy regimen in the metastatic setting
* Measurable disease by RECIST Criteria

Exclusion Criteria:

* Received prior lapatinib, an investigational ErbB-2 and/or an investigational EGFR dual tyrosine kinase inhibitors
* Administration of any other chemotherapy, biological, immunotherapy or investigational agent within 14 days prior to receipt of study medication
* Pregnant or breast-feeding women. Known CNS metastases, unless treated and without clinically significant neurological deficits
* Moderately severe dry eye
* Congestive heart failure, or a left ventricular ejection fraction
* Myocardial infarction or active ischemic heart disease within 12 months prior to study drug administration
* Previous malignancies unless free of recurrence for at least 5 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-04; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Objective tumor response rate (either RECIST or WHO complete response, partial response or minor response) confirmed by CT and MRI as the preferred methods for tumor assessments and Chest x-ray is acceptable for pulmonary lesions | Within 28 days prior to the start of treatment with tumor assessments reevaluated every 8 weeks (+/- 4 days)
  (all patients were off study by June 2008)

SECONDARY OUTCOMES:
Adverse Events assessed according to the NCI CTCAE (v 3.0) grading system | Within 28 days prior to the start of treatment, and for 167 days
  (all patients were off study by June 2008)
Laboratory tests assessed according to the NCI CTCAE (v 3.0) grading system | Within 10 days prior to Cycle 1/1st infusion; within 48 hours of infusion (Cycle 1/Weeks 2/3/4 and Cycle 2+/Week3), or within 72 hours prior to infusion (Cycle 2+/Week 1)
Vital signs | Within 28 days prior to the start of treatment, Day1 of Weeks 1, 2, and 3 of Cycle 1 (4 weeks long), and prior to each 4-week cycle starting with Cycle 2, for 167 days
  (all patients were off study by June 2008)
Karnofsky Performance Status | Within 28 days prior to the start of treatment, prior to each 4-week cycle starting with Cycle 2, for 167 days
  (all patients were off study by June 2008)
Ocular testing | Within 28 days prior to the start of treatment, Cycle 1/Day 10 (3 days +/- 1 day following the 2nd infusion in the first cycle of therapy), prior to Cycle 2, if clinically indicated thereafter, for 167 days
  (all patients were off study by June 2008)
Kaplan-Meier estimate of time to progression | Within 28 days prior to the start of treatment with tumor assessments reevaluated every 8 weeks (+/- 4 days)
  (all patients were off study by June 2008)
Time to progression on the patient's prior cytotoxic chemotherapy compared to the patient's time to progression on alvespimycin | Within 28 days prior to the start of treatment with tumor assessments reevaluated every 8 weeks (+/- 4 days)
  (all patients were off study by June 2008)
Kaplan-Meier estimate of progression-free survival | Within 28 days prior to the start of treatment with tumor assessments reevaluated every 8 weeks (+/- 4 days)
  (all patients were off study by June 2008)
Kaplan-Meier estimate of time to response | Within 28 days prior to the start of treatment with tumor assessments reevaluated every 8 weeks (+/- 4 days)
  (all patients were off study by June 2008)
Kaplan-Meier estimate of duration of response | Within 28 days prior to the start of treatment with tumor assessments reevaluated every 8 weeks (+/- 4 days)
  (all patients were off study by June 2008)
Kaplan-Meier estimate of time to treatment failure | Within 28 days prior to the start of treatment with tumor assessments reevaluated every 8 weeks (+/- 4 days)
  (all patients were off study by June 2008)
Kaplan-Meier estimate of overall survival | Within 28 days prior to the start of treatment with tumor assessments reevaluated every 8 weeks (+/- 4 days)
  (all patients were off study by June 2008)
Changes in tumor markers | Within 28 days prior to the start of treatment, Prior to each 4-week cycle starting with Cycle 2, for 167 days
Histopathological and molecular profile of responding and non-responding patients using paraffin-embedded surgical specimens | Specimens were obtained within 28 days prior to the start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb